CLINICAL TRIAL: NCT03926299
Title: Prospective, Randomized, Active-controlled Investigator Initiated Clinical Trial to Demonstrate That the Nd:YAG/Er:YAG Dual Laser Therapy is Effective to Treat Vulvar Lichen Sclerosus and Similar to Standard Treatment With Steroid Cream
Brief Title: Clinical Trial to Demonstrate That the Dual Laser Therapy is Effective for the Treatment of Vulvar Lichen Sclerosus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Volker Viereck (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Volker Viereck, Head of Urogynecology, Cantonal Hospital, Frauenfeld
Organization: Cantonal Hospital, Frauenfeld (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lichen sclerosus laser study
Record Dates: First submitted 2019-04-18; First posted 2019-04-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Chronic Skin Disease; Vulvar Lichen Sclerosus
MeSH Terms: conditions — Vulvar Lichen Sclerosus | interventions — Laser Therapy; Clobetasol; Ointments

STUDY DESIGN:
Intervention Model Description: randomized, active-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser (Experimental): dual Fotona laser treatment (Nd:YAG and Er:YAG)
  Interventions: Device: FotonaSmooth SP® Spectro laser device
- Topical steroid (Active Comparator): clobetasol propionate 0.05% cream
  Interventions: Drug: Clobetasol propionate 0.05% ointment

INTERVENTIONS:
Device: FotonaSmooth SP® Spectro laser device — dual laser treatment with thermal Nd:YAG and ablative Er:YAG (Fotona medical device), 4 laser sessions 4-8 weeks apart.
  Other Names: Laser therapy
  Arms: Laser
Drug: Clobetasol propionate 0.05% ointment — 6 months standard treatment with topical steroid cream (high dose for the first two months, medium dose for the next two months, low dose for the last two months)
  Other Names: Local steroid therapy
  Arms: Topical steroid

SUMMARY:
The aim of this study is to test a new, minimally invasive dual laser technique to treat vulvar lichen sclerosus. Efficacy and safety of the thermal non-ablative Nd:YAG laser and the ablative Er:YAG laser is determined and compared to the current standard treatment with high dose steroids. The hypothesis is that laser therapy is effective and similar to standard steroid therapy.

DETAILED DESCRIPTION:
Lichen sclerosus (LS) is a chronic inflammatory skin disease that usually involves the anogenital area where it causes itching and burning pain, pain during sexual intercourse, and anal or genital bleeding due to fissuring of the damaged tissue. In this study a treatment with dual laser application combining thermal non-ablative Nd:YAG with ablative Er:YAG laser is used to reduce the symptoms of LS. Results will be compared to the standard therapy with topical steroid cream.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of vulvar lichen sclerosus
* Clinical LS score ≥ 4

Exclusion criteria:

* Concomitant steroid, calcineurin inhibitor or any other topical or systemic treatment for LS
* < 3 months since start of vaginal estrogen treatment
* Malignant disease as the cause of the vulval symptoms
* BMI > 35 kg/m²
* Acute infection (fungal, bacterial, viral) of the vulva, vagina or bladder
* Presence of contraindications for the laser treatment or topical steroid treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Lichen sclerosus score (LS score) | 6 months
  Reduction (i.e. improvement) of physician administered clinical LS score (Sum score of 6 items on a scale from 0-2 (0=no, 1=weak, 2=pronounced): erosions, hyperkeratosis, fissures, agglutination, stenosis, atrophy). Possible sum score ranges from 0 (normal) to 12 (maximum symptoms present).

SECONDARY OUTCOMES:
Vulvovaginal symptom questionnaire (VSQ) | At each visit through study completion, an average of 1 year
  21 binary questions (0=no, 1=yes) about symptoms, emotional impact, impact on quality of life, impact on sexual activity. Total possible sum score is 21.
Symptom strength score | At each visit through study completion, an average of 1 year
  Visual analog scale (0-10) of LS symptoms itching, burning, vulvar pain, dyspareunia. Total sum score ranges from 0 (no symptoms) to 40 (maximal symptoms).

OTHER OUTCOMES:
Vulvar punch biopsy | Baseline and at 6 months
  Histological changes
Photo documentation of vulvar skin | At each visit through study completion, an average of 1 year
  Changes of visual appearance of vulvar skin
Patient satisfaction | At each follow-up visit (6 months and 12 months)
  Satisfaction of the treatment. Levels: 3 = very much better, 2 = much better, 1 = a little better, 0 = no change, -1 = a little worse, -2 = much worse, -3 = very much worse
Pain during treatment (for laser arm only): Visual analog scale (0-10) | At each laser treatment session (baseline, 1 month, 2 months, 4 months)
  Visual analog scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Volker Viereck, Prof., Principal Investigator — Department of Gynecology and Obstetrics
Locations (1):
- Cantonal Hospital Frauenfeld, Frauenfeld, Thurgau, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zivanovic I, Gamper M, Fesslmeier D, Bischofberger H, Viereck V. A randomized controlled trial to evaluate a novel dual laser therapy for vulvar lichen sclerosus: exploratory study assessing the impact of menopausal status. Menopause. 2025 Mar 1;32(3):228-233. doi: 10.1097/GME.0000000000002478. Epub 2025 Feb 21. PMID 39998969
- [Derived] Viereck V, Gamper M, Regauer S, Walser C, Zivanovic I. Nd:YAG/Er:YAG dual laser vs. topical steroid to treat vulvar lichen sclerosus: study protocol of a randomized controlled trial. Arch Gynecol Obstet. 2023 Aug;308(2):643-649. doi: 10.1007/s00404-023-07055-z. Epub 2023 May 5. PMID 37145134